CLINICAL TRIAL: NCT06058728
Title: A Prospective, Single-Arm, Descriptive Observational Study to Evaluate Changes in Hair in Women Exposed to Oriahnn® (Elagolix 300 mg BID With Estradiol 1 mg/Norethindrone Acetate 0.5 mg QD)
Brief Title: A Study to Evaluate Changes in Hair in Adult Participants Taking Oral Oriahnn Capsules With Heavy Menstrual Bleeding (HMB) Associated With Uterine Fibroids (UF)
Acronym: Pink Orchid
Status: Withdrawn | Type: Observational
Why Stopped: Company Decision
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P20-400
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Uterine Fibroids (UF)
Keywords: Uterine Fibroids (UF); Heavy Menstrual Bleeding (HMB); Oriahnn; Elagolix; Estradiol; Norethindrone Acetate
MeSH Terms: conditions — Leiomyoma; Menorrhagia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Part 1 - Oriahnn Exposure Cohort: Participants prescribed Oriahnn for management of heavy menstrual bleeding (HMB) due to uterine fibroids (UF).
- Part 2 - Nested Hair Loss Cohort: Participants prescribed Oriahnn for management of HMB due to UF, with meaningful hair loss.

SUMMARY:
Uterine Fibroids (UF) are benign smooth muscle neoplasms of the uterus that affect women of reproductive age. UFs are one of the leading causes of hospitalizations for gynecological disorders and often lead to hysterectomy. In this study, women with heavy menstrual bleeding (HMB) due to UF who are being treated with Oriahnn will be followed to establish the incidence rate, time to onset, extent, pattern, and resolution of meaningful hair loss, as well as any racial differences.

Oriahnn is an approved drug for the management of HMB associated with UF. All study participants will receive Oriahnn as prescribed by their study doctor in accordance with approved local label. Study Participants will be followed for up 24 months (part 1). Approximately 1600 participants aged 18-50 years will be enrolled at 1 site in the United States.

Participants will receive oral Oriahnn as prescribed by their physician according to their routine clinical practice and local label. Participants will be followed for 24 months.

There is expected to be no additional burden for participants in this trial. Participants will complete questionnaires on a quarterly basis.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

* International Classification of Disease-10 (ICD-10) diagnosis codes for both uterine fibroids (UF) (D25.X) and heavy menstrual bleeding (HMB), defined as menorrhagia (N92.0, N92.4) or menometrorrhagia (N92.1) in the electronic health record (EHR) system.
* Plans to initiate or has initiated Oriahnn treatment within 14 days of study enrollment.
* Able to provide photographs of their scalp within 14 days of Oriahnn initiation, based on instruction provided.

Part 2:

- Changes in thickness, fullness or pattern of hair that results in less hair than normal, or hair shedding that is increased from normal in the Hair Questionnaire.

Exclusion Criteria:

* Current or history of hair thinning, hair loss, or alopecia (defined as physician-diagnosed or patient-reported hair loss).
* Have a contraindication to receive Oriahnn per Prescribing Information.
* Any of the following occurrences within 180 days prior to Oriahnn prescription.

  * Prescription for Oriahnn, another gonadotropin releasing hormone (GnRH) antagonist [including Myfembree (relugolix, estradiol/norethindrone acetate]) or GnRH agonist.
  * Pregnancy/Childbirth.
  * New diagnosis of thyroid disease.
  * New diagnosis of inflammation or infection of the scalp (e.g., psoriasis, tinea capitis).
  * Have taken medications or undergone therapies that may cause alopecia, hair loss, or both. This includes but is not limited to chemotherapy, checkpoint inhibitors, epidermal growth factor antagonists, or radiation anywhere on the body.
* Initiation or changes in medications or doses for the management of thyroid diseases
* Any other medical condition or surgery requiring hospitalization (other than UF)

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women 18 to 50 years old with heavy menstrual bleeding (HMB) due to uterine fibroids (UF).
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Meaningful Hair Loss | Up to Month 24
  Meaningful hair loss is defined as patient-reported changes in thickness, fullness, or pattern of hair that results in less hair than normal or hair shedding that is increased from normal in the Hair Questionnaire.
Time to Onset of Hair Loss | Up to Month 42
  Time from initiation of Oriahnn until patient-reported meaningful hair loss will be assessed.
Changes in Patterns of Hair Loss | Up to Month 42
  Based on example description and images of alopecia subtypes, changes in patterns of hair loss are classified as primary pattern of hair loss.
Number of Participants with Improvement in Hair Loss | Up to Month 42
  Defined as a report that since the participant has reported hair loss, her hair loss has improved.
Number of Participants with Resolution in Hair Loss | Up to Month 42
  Resolution in hair loss is defined as a report that since the patient has reported hair loss, her hair has returned to normal.
Time to Resolution in Hair Loss | Up to Month 42
  Time from onset of meaningful hair loss until reported resolution.
Number of Participants who Discontinued Oriahnn at Reported Hair Loss | Up to Month 42
  Discontinuations of Oriahnn at or after reported hair loss will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (1):
- Dorsata /ID# 252675, Arlington, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P20-400